CLINICAL TRIAL: NCT06807203
Title: Spontaneous Motor-voice Assessment in Infants Using Video and Audio Recordings.
Brief Title: Motor-voice Assessment in Infants (MAMI)
Acronym: MAMI
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jill Heathcock, Professor, Ohio State University
Other Study IDs: 2024B0149
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy Infantile; Pre-Term; Motor Delay; Neurodevelopmental Disorders; Autism Spectrum Disorder
Keywords: Digital health,; Motor assessment,; voice assessment,; cognition; neurodevelopment,
MeSH Terms: conditions — Cerebral Palsy; Premature Birth; Psychomotor Disorders; Neurodevelopmental Disorders; Autism Spectrum Disorder | interventions — Behavior Observation Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Full-term and pre-term infants: Observational study for motor, cognitive, language, voice impairments.
  Interventions: Other: Behavioral observation

INTERVENTIONS:
Other: Behavioral observation — Behaviors will be observed in children's natural environment. With a digital health assessment.

SUMMARY:
The goal of this observational study is to discover features of normal and disordered motor-voice profiles that are biobehavioral markers of physical disability in infants.. The main questions it aims to answer are:

Identify voice factors among infants with newborn-detectable risk. Identify association between individual characteristics (Gestational age at birth, global function, motor-function) and voice factors.

Examine unique features of voice production that are present in infants with high-risk for Cerebral Palsy (CP).

Participants will be asked to upload a 3-minute videos of their child at term-age, 3.5-, and 9-months of age.

At the 3.5-month and 9-month time point parents can choose to attend an optional in-person assessment with their child.

DETAILED DESCRIPTION:
In the first months of life, infants continually produce and modify motor behaviors and acquire new ones. They kick their legs in patterns that show temporal and spatial organization, they flap their arms in a march to midline, and gain strength against gravity with their head and trunk. Most of this happens spontaneously without specific toys or environmental modifications. Over the same time period, infant also continually use and modify their voice and acquire new vocal behaviors. Three broad categories of sound occurring in vocal communication are described in infants: cries, laughs, and protophones which are seen as the precursors to speech. Motor function and voice production are not isolated developmental processes --they are present and developing in the same baby, and, they have common ontological origins in the motor cortex. It can be argued that the earliest precursors to language, spontaneous cries and protophones, are the result of a "movement" originating in signals from the CNS that can be studied to detect health and disease in combination with physical movements. Grounded in the developmental cascades framework and developmental neuroscience this project is informed by clinical and scientific advancements in: 1) Methodology for reliably scoring of spontaneous behaviors in the first months of life that are sensitive to normal and disordered movements and predictive of neurodevelopmental disabilities including Cerebral Palsy (CP) - particularly the General Movements Assessment (GMA) and associated Motor Optimality score (MOS); 2) The ability to detect abnormal voice production in populations with neurodevelopmental disabilities using acoustic analysis. Motor function and speech production are complex processes that require precise coordination of 100s of muscles. In disease states, with damage to the CNS, poor coordination can be observed through motor and voice behaviors and specific diseases identified. Importantly, motor and voice are some of the first indicators of health after birth that occur spontaneously (e.g. crying, kicking, muscle tone). Even more importantly, motor function and voice production can be measured, non-invasively, in early infancy including the newborn period.

The overall goal is to discover features of normal and disordered motor-voice profiles that are biobehavioral markers of physical disability in infants. Disabilities are difficult to identify in this ultra-early infancy period because infants cannot speak or produce voluntary movements necessary for formal testing. Furthermore, medical testing such as MRI is expensive, not accessible everywhere, and has limited predictive value for neurodevelopmental outcomes. Laboratories have demonstrated the promise of using video and audio recordings from spontaneous and elicited behaviors to identify disordered motor or voice production from normal. Arm and leg movements, midline behaviors, writhing and fidgety movements are all implicated in neurodevelopmental outcomes and some are uniquely implicated in the identification of cerebral palsy (CP). Vocalizations (grunts, squeals, raspberries, trills, clicks), crying, protophones -- core behavioral features of voice production, are also implicated in neurodevelopmental outcomes; and some are uniquely implicated in autism, but none have been consistently evaluated in infants. Multidimensional assessment of motor function and voice production will be used at two time periods that are relevant to the earliest possible screening and detection of neurodevelopmental disorders and important for general movement assessment: term-equivalent age (writhing period), 3.5 months of corrected age (fidgety period), and 9 month of corrected age in N=46 infants with newborn-detectable risk. To fully capture the complexity of motor function and voice production in infancy, a battery of tests with emerging sensitivity will be used to measure disability during development and the sensitivity to detect both major impairments and small delays; some of these measures can be reliably tested simultaneously. Tests include: (1) General Movement Analysis (GMA); (2) the GMA-associated Motor Optimality Score (MOS); (3) Voice acoustic analysis (fundamental frequency, ratio of voiced sound, shimmer, jitter, Harmonic-to-noise ratio, frequencies of the first four formants), and number of vocalizations; (4) Bayley Scales of Infant Development (Bayley-4) for motor, cognitive, and language function; (5) Test of Infant Motor Performance (TIMP); and (6) Ages and Stages Questionnaire (ASQ).

ELIGIBILITY:
Inclusion Criteria:

* gestational age of 24 0/7 - 41 6/7,
* admitted to the NICU,
* medically stable by 40 weeks of gestation (including off ventilator support),
* born to mothers 18 - 43 years old at the time of birth,
* one parent fluent in English.

Exclusion Criteria:

* diagnosis of a genetic syndrome (e.g. Trisomy 21),
* musculoskeletal deformity,
* failed hearing screen.

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Full-term and pre-term infants
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2028-01-28 (Estimated); Study Completion 2030-01-28 (Estimated)

PRIMARY OUTCOMES:
General Movement Assessment | At term-age, 3- and 9-months corrected age.
  A non-invasive medical exam that evaluates an infant's spontaneous movements to identify neurological issues.
GMA-associated Motor Optimality Score | At term-age, 3- and 9-months corrected age.
  A numerical score derived from the General Movements Assessment (GMA), a method used to evaluate an infant's spontaneous movements, where a higher score indicates more optimal motor development and a lower score may suggest potential neurological concerns.
Voice acoustic analysis and number of vocalizations | At term-age, 3- and 9-months corrected age.
  Fundamental frequency, ratio of voiced sound, shimmer, jitter, Harmonic-to-noise ratio, frequencies of the first four formants

SECONDARY OUTCOMES:
Ages and Stages Questionnaire | 3- and 9-months corrected age.
  Screens children from birth to six years old for developmental and social-emotional progress.
Bayley Scales of Infant Development | Optional at 3.5- and 9-months corrected age.
  Comprehensive assessment tool for determining developmental delays in children. Scores are given as polytomous, ranging from 0 to 2. Scoring: 2 are Mastery, 1 is emerging, and 0 means absent. Mean score of 100 (Standard Deviation=15) at the 50th percentile signifies mid-average functioning. Scores below 85 (1 Standard Deviation below the mean), at the 16th percentile, indicate mild impairment of being 'at risk' of developmental delay.
Test of Infant Motor Performance | Optional at 3.5- and 9-months corrected age.
  A 42-item assessment that measures an infant's motor skills and posture.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States